CLINICAL TRIAL: NCT00819234
Title: Extension Study of Protocol DFA102 to Examine the Long-Term Safety, Tolerability, and Effect on Body Weight of Pramlintide Administered in Combination With Metreleptin in Obese and Overweight Subjects
Brief Title: Extension Study of Protocol DFA102 to Examine the Long-Term Safety, Tolerability, and Effect on Body Weight of Pramlintide Administered in Combination With Metreleptin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFA102E
Record Dates: First submitted 2008-12-24; First posted 2009-01-08 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Leptin; Pramlintide; Obese; Symlin; Amylin
MeSH Terms: conditions — Obesity | interventions — pramlintide; metreleptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental): Pramlintide and 1.25mg Metreleptin
  Interventions: Drug: Pramlintide and Metreleptin
- 3 (Experimental): Pramlintide and 2.5mg Metreleptin
  Interventions: Drug: Pramlintide and Metreleptin
- 4 (Experimental): Pramlintide and 5.0mg Metreleptin
  Interventions: Drug: Pramlintide and Metreleptin

INTERVENTIONS:
Drug: Placebo — placebo pramlintide and placebo metreleptin twice daily
  Arms: 1
Drug: Pramlintide and Metreleptin — Subcutaneous injection, twice daily
  Other Names: Symlin
  Arms: 2; 3; 4

SUMMARY:
Study DFA102E is an extension of Study DFA102, which included a 28-week treatment period with randomized study medication. The purpose of the extension study is to examine the long-term (up to 1 year) safety, tolerability, and effect on body weight of treatment with pramlintide and metreleptin, administered as separate subcutaneous (SC) injections, in obese and overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study DFA102, including all procedures required at the Study Termination visit, without major protocol deviations
* Male, or female and meets all the following criteria:

  1. Has a negative urine pregnancy test result at Study start(not applicable to hysterectomized females)
  2. If of childbearing potential must practice and be willing to continue to practice appropriate birth control during the entire duration of the study
* Able to read, understand, and sign the Informed Consent Form (ICF) and if applicable,an Authorization to Use and Disclose Protected Health Information Form, answer the study questionnaires, communicate with the investigator, and understand and comply with protocol requirements

Exclusion Criteria:

* Is expected to require or undergo treatment with any exclusionary medication.
* Is undesirable as a study participant as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Chan, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (33):
- United States (33):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arkansas
  - Research Site, Santa Rosa, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Plantation, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Edina, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Anderson, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Olympia, Washington

REFERENCES:
- [Derived] Chan JL, Koda J, Heilig JS, Cochran EK, Gorden P, Oral EA, Brown RJ. Immunogenicity associated with metreleptin treatment in patients with obesity or lipodystrophy. Clin Endocrinol (Oxf). 2016 Jul;85(1):137-49. doi: 10.1111/cen.12980. Epub 2016 Feb 2. PMID 26589105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (overweight and obese) must have been randomized and treated in original DFA102 Study (NCT00673387) in order to be enrolled into this extension study DFA102E and followed for a total of up to 52 weeks, inclusive of DFA102 (ie, DFA102 and DFA102E studies together have a total length of 52 weeks).
Pre-assignment Details: DFA102 participants assigned to: placebo, 360mcg pramlintide+1.25mg metreleptin, 360mcg pram+2.5mg metre, or 360mcg pram+5.0mg metre did not change treatment in extension (stable groups). All other groups transitioned to 360mcg pram + 1.25, 2.5 or 5.0mg metre. 274 enrolled in extension and 273 were treated.
Groups:
- Placebo - Stable: Placebo matched to pramlintide BID plus placebo matched to metreleptin BID self administered subcutaneously (SC) for 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E.
- 360 mcg Pramlintide + 1.25mg Metreleptin - Stable: Participants who received 360 mcg pramlintide plus 1.25 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
- 360 mcg Pramlintide + 2.5 Metreleptin - Stable: Participants who received 360 mcg pramlintide plus 2.5 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
- 360 mcg Pramlintide + 5.0 Metreleptin - Stable: Participants who received 360 mcg pramlintide plus 5.0 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E.
- 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Monotherapy: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 1.25 metreleptin in this group of the extension study for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Monotherapy: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 2.5 metreleptin in this group of the extension study for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Monotherapy: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 5.0 metreleptin in this group of the extension study for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono: Participants who received 5.0 mg metreleptin plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 5.0 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102. A blinded pramlintide dose escalation/titration in the first week of treatment was performed for participants who had not received 360 mcg pramlintide in DFA102, to minimize nausea and/or vomiting.
- 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram: Participants who received 180 mcg pramlintide plus 2.5 mg metreleptin self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg pramlintide plus 2.5 mg metreleptin in the extension study for up to 52 Weeks, inclusive of DFA102. A blinded pramlintide dose escalation/titration in the first week of treatment was performed for participants who received 180 mcg pramlintide in DFA102, to minimize nausea and/or vomiting.
- 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram: Participants who received 180 mcg pramlintide plus 5.0 mg metreleptin self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg pramlintide plus 5.0 mg metreleptin in the extension study for up to 52 Weeks, inclusive of DFA102. A blinded pramlintide dose escalation/titration in the first week of treatment was performed for participants who received 180 mcg pramlintide in DFA102, to minimize nausea and/or vomiting.
Period: Overall Study
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Monotherapy | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Monotherapy | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Monotherapy | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Started | 31 | 35 | 36 | 28 | 13 | 14 | 13 | 29 | 37 | 37
Completed | 21 | 20 | 28 | 22 | 12 | 7 | 8 | 20 | 31 | 30
Not Completed | 10 | 15 | 8 | 6 | 1 | 7 | 5 | 9 | 6 | 7
Not completed — Withdrawal by Subject | 8 | 13 | 6 | 3 | 0 | 4 | 4 | 8 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who completed original study and chose to be enrolled into this extension study and were treated with study drug.
Groups:
- All Participants: All participants who completed the original study and chose to enter the extension study.
Arm/Group | All Participants
Number analyzed (Participants) | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191
  Male | 82
Region of Enrollment [Number; unit: participants]
  United States | 273
Body Weight at Baseline [Mean (Standard Deviation); unit: kilograms] — Baseline in the extension study was Week 28 in the original study. If Week 28 value was missing or after the first dose in DFA102E, the last available value on or prior to Week 28 was used.
  kilograms | 95.83 (17.007)
Body Mass Index (BMI) at Baseline [Mean (Standard Deviation); unit: kg/m^2] — Baseline refers to Week 28 in original study. If Week 28 was missing or after the first dose in DFA102E, the last available value on or prior to Week 28 was used. Body Mass Index (BMI) was measured as kilogram per meter of height squared (kg/m^2).
  kg/m^2 | 34.16 (4.988)

OUTCOME MEASURES:

1. Primary Outcome: LS Mean Percent Change in Body Weight From Original Study DFA102 (NCT00673387) Baseline (Day 1) at Week 52 in Extension Study DFA102E - Evaluable Treatment Stable Population
Description: Original study DFA102 (NCT00673387) baseline refers to Visit 5 (Day 1). If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Least Squares (LS) Mean based on a repeated measures mixed model with treatment, sex, DFA102 baseline BMI category, nominal week, treatment by nominal week interaction as factors, and DFA102 baseline weight value as a covariate, with a heterogeneous compound symmetry error covariance structure within each treatment group. Stable population consists of all ITT participants (received at least one injection of treatment) who had the same treatment group assignment in Study DFA102 and Study DFA102E, ie, ITT participants who were in Study DFA102 treatment groups Placebo, Pramlintide 360 + Metreleptin 1.25, Pramlintide 360 + Metreleptin 2.5 and Pramlintide 360 + Metreleptin 5.0.
Time Frame: Original Study Baseline to Week 52
Population: Enrolled and received at least 1 injection of any treatment (ITT); treatment regimens same in both DFA102/DFA102E (stable); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock); no major deviations during original study/extension. Additional exclusions based on clinical review of the data prior database lock.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in weight
Groups:
- Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 1.25 mg BID self administered SC. All participants entered treatment for 52 Weeks, inclusive of DFA102.
- Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 2.5 mg BID self administered SC. All participants entered treatment for 52 Weeks, inclusive of DFA102.
- Pramlintide 360 Mcg + Metreleptin 5.0 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 5.0 mg BID self administered SC for 52 Weeks, inclusive of DFA102.
Arm/Group | Placebo - Stable | Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable | Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable | Pramlintide 360 Mcg + Metreleptin 5.0 mg - Stable
Number analyzed (Participants) | 21 | 20 | 27 | 19
percentage of change in weight | -2.68 (2.170) [-7.00 to 1.64] | -9.92 (2.203) [-14.30 to -5.53] | -9.24 (1.944) [-13.10 to -5.37] | -8.20 (2.201) [-12.58 to -3.82]
Statistical Analysis 1: Comparison: Placebo - Stable vs Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable; Treatment comparisons between each active treatment and placebo. Statistical tests performed two-sided at a significance level of α = 0.05. The null hypothesis tested was that there is no difference between each active treatment and the placebo treatment. The primary analysis did not incorporate any adjustment for multiple comparisons; Test type: Superiority or Other; p = 0.0135, t-test, 2 sided; LS Mean Difference = -7.23, 95% CI 2-sided [-12.93 to -1.54], Standard Error of Mean 2.863
Statistical Analysis 2: Comparison: Placebo - Stable vs Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0168, t-test, 2 sided; LS Mean = -6.55, 95% CI 2-sided [-11.89 to -1.21], Standard Error of Mean 2.681
Statistical Analysis 3: Comparison: Placebo - Stable vs Pramlintide 360 Mcg + Metreleptin 5.0 mg - Stable; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0595, t-test, 2 sided; LS Mean = -5.52, 95% CI 2-sided [-11.27 to 0.23], Standard Error of Mean 2.887

2. Secondary Outcome: LS Mean Absolute Change in Body Weight From Original Study Baseline (Day 1) at Weeks 12, 28, 36, 44, and 52 - Evaluable Treatment Stable Population
Description: Original study DFA102 (NCT00673387) baseline refers to Visit 5 (Day 1). If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Weeks 12 and 28 were in original study (Week 28 was baseline for extension study), while Weeks 36, 44, and 52 were in the extension study. Body weight was measured in kilograms (kg).
Time Frame: Original baseline to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Groups:
- Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 1.25 mg BID self administered SC for 52 Weeks, inclusive of DFA102.
- Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 2.5 mg BID self administered SC for 52 Weeks, inclusive of DFA102.
Arm/Group | Placebo - Stable | Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable | Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable | Pramlintide 360 Mcg + Metreleptin 5.0 mg - Stable
Number analyzed (Participants) | 31 | 35 | 36 | 28
kg
  Week 12 (original study) | -4.59 [-6.55 to -2.62] | -6.72 [-8.71 to -4.73] | -7.31 [-9.07 to -5.55] | -7.06 [-9.05 to -5.07]
  Week 28 (Baseline for Extension) | -3.70 [-6.74 to -0.66] | -8.63 [-11.72 to -5.55] | -9.91 [-12.64 to -7.19] | -9.46 [-12.55 to -6.38]
  Week 36 in Extension Study | -3.53 [-6.95 to -0.12] | -9.74 [-13.21 to -6.27] | -10.69 [-13.75 to -7.63] | -9.21 [-12.68 to -5.75]
  Week 44 in Extension Study | -3.10 [-6.82 to 0.63] | -9.38 [-13.16 to -5.60] | -10.00 [-13.33 to -6.66] | -8.60 [-12.38 to -4.82]
  Week 52 in Extension Study | -2.85 [-6.98 to 1.28] | -9.26 [-13.45 to -5.07] | -9.65 [-13.35 to -5.96] | -7.98 [-12.16 to -3.79]

3. Secondary Outcome: Fasting Total Leptin Concentration by Visit and Pooled Metreleptin Stable Treatment by Metreleptin Dose - Week 52 Stable Evaluable Population
Description: Baseline is Day 1 in original study DFA102, baseline in DFA102E is Week 28. Follow up is 3 - 28 days after the end of treatment period. As total leptin is measured, placebo arm was not included in the evaluation. Fasting total leptin is measured in nanograms per milliliter (ng/mL). The assay for measuring total plasma leptin is not specific for metreleptin and detects both endogenous leptin and exogenous metreleptin.
Time Frame: Original Study Baseline to Extension Week 52 and follow up
Population: Enrolled and received at least 1 injection of metreleptin; treatment regimens same in both DFA102/DFA102E (stable population); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock); no major deviations during original study/extension.
Measure: Geometric Mean (Standard Error); unit: ng/mL
Groups:
- Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 1.25 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
- Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 2.5 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
- Pramlintide 360 Mcg + Metreleptin 5.0 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 5.0 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
Arm/Group | Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable | Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable | Pramlintide 360 Mcg + Metreleptin 5.0 mg - Stable
Number analyzed (Participants) | 20 | 27 | 19
ng/mL
  DFA102 Baseline | 32.50 (4.990) | 34.48 (3.089) | 29.50 (2.251)
  DFA102E Baseline (Week 28) | 102.02 (17.466) | 232.48 (29.371) | 420.24 (48.012)
  Week 40 | 96.23 (19.418) | 236.02 (29.856) | 416.52 (58.352)
  Week 52 | 88.47 (17.576) | 177.32 (25.765) | 259.85 (40.650)
  Follow up post treatment | 52.90 (9.584) | 89.21 (11.180) | 89.49 (11.712)

4. Secondary Outcome: LS Mean Absolute Change in Waist Circumference From Baseline in the Original Study to Week 52 in the Extension Study - Week 52 Evaluable Stable Population
Description: Baseline is the baseline in the original study DFA102 (Day 1). If Day 1 value was missing or after the first dose of drug, the last available value on or prior to Day 1 was used. Waist circumference was measured in centimeters (cm). Week 52, treatment stable evaluable population: those participants who enrolled and received at least 1 injection of any treatment (ITT); treatment regimens same in both DFA102/DFA102E (stable); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock); no major deviations during original study/extension. Additional exclusions based on clinical review of the data prior database lock.
Time Frame: Baseline to Week 52
Population: n=number of participants with non-missing waist circumference data at this visit in each treatment group. Week 12 n=21,20,27,19; Week 28 n=21,20,26,19; Week 36 n=21,20,27,19; Week 44 n=20,20,27,19; Week 52 n=21,19,27,19.ITT population with treatment regimens same in DFA102/DFA102E; completed Week 52; no major protocol deviations in DFA102/102E.
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Groups:
- Placebo: Placebo matched to pramlintide BID plus placebo matched to metreleptin BID self administered subcutaneously (SC) for 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 1.25mg Metreleptin - Stable: Participants who received 360 mcg pramlintide plus 1.25 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 2.5 Metreleptin - Stable: Participants who received 360 mcg pramlintide plus 2.5 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 5.0 Metreleptin - Stable: Participants who received 360 mcg pramlintide plus 5.0 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
Arm/Group | Placebo | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable
Number analyzed (Participants) | 21 | 20 | 27 | 19
cm
  Week 12 (original study) | -4.62 [-7.15 to -2.08] | -4.03 [-6.57 to -1.49] | -5.77 [-8.03 to -3.51] | -5.70 [-8.25 to -3.15]
  Week 28 (baseline in Extension study) | -3.37 [-6.63 to -0.10] | -6.48 [-9.75 to -3.20] | -7.95 [-10.92 to -4.97] | -8.36 [-11.65 to -5.07]
  Week 36 Extension study | -3.24 [-6.77 to 0.29] | -8.79 [-12.33 to -5.25] | -9.19 [-12.34 to -6.04] | -8.16 [-11.71 to -4.60]
  Week 44 Extension study | -3.46 [-7.20 to 0.28] | -9.09 [-12.74 to -5.44] | -9.03 [-12.27 to -5.78] | -8.76 [-12.42 to -5.10]
  Week 52 Extension study | -3.69 [-7.43 to 0.05] | -9.08 [-12.95 to -5.21] | -9.18 [-12.52 to -5.84] | -7.41 [-11.18 to -3.65]

5. Secondary Outcome: LS Mean Percent Change in Body Weight From Baseline of Original Study DFA102 at Week 12, and at Weeks 28, 36, 44, and 52 in the Extension Study DFA102E - Week 52 Evaluable Treatment Stable Population
Description: Baseline is Day 1 in study DFA102. If Day 1 value was missing or after the first dose of drug, the last available value on or prior to Day 1 was used. Baseline in the Extension Study was Week 28. Week 52, treatment stable evaluable population: those participants who enrolled and received at least 1 injection of any treatment (ITT); treatment regimens same in both DFA102/DFA102E (stable); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock).
Time Frame: Baseline to Week 52
Population: n=number of participants with non-missing data at this visit in each treatment group. Week 12 n=21,20,27,19; Week 28 n=21,20,27,19; Week 36 n=21,20,27,19; Week 44 n=21,20,27,19; Week 52 n=21,20,27,19. ITT population with treatment regimens same in DFA102/DFA102E; completed Week 52; no major protocol deviations in DFA102/102E.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change in weight
Groups:
- Placebo - Stable: Placebo matched to pramlintide BID plus placebo matched to metreleptin BID self administered subcutaneously (SC) for 52 Weeks, inclusive of DFA102.
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable
Number analyzed (Participants) | 21 | 20 | 27 | 19
Percentage of change in weight
  Week 12 of original study | -4.56 [-6.48 to -2.65] | -6.93 [-8.87 to -4.99] | -7.23 [-8.95 to -5.52] | -7.17 [-9.11 to -5.23]
  Week 28 Extension study | -3.78 [-6.83 to -0.74] | -9.14 [-12.22 to -6.05] | -9.72 [-12.44 to -6.99] | -9.83 [-12.91 to -6.74]
  Week 36 Extension study | -3.43 [-6.91 to 0.05] | -10.27 [-13.80 to -6.74] | -10.43 [-13.55 to -7.32] | -9.51 [-13.04 to -5.98]
  Week 44 Extension study | -3.01 [-6.86 to 0.84] | -9.95 [-13.86 to -6.04] | -9.65 [-13.09 to -6.20] | -8.84 [-12.75 to -4.94]
  Week 52 Extension study | -2.68 [-7.00 to 1.64] | -9.92 [-14.30 to -5.53] | -9.24 [-13.10 to -5.37] | -8.20 [-12.58 to -3.82]

6. Secondary Outcome: LS Mean Absolute Change From Baseline in Original Study DFA102 to Week 52 in Extension Study DFA102E for Glucose and Lipids - Week 52 Evaluable Treatment Stable Population
Description: Glucose, total cholesterol, triglycerides, low density lipoprotein (LDL), and high density lipoprotein (HDL) were measured in milligrams per deciliter (mg/dL). Baseline was Day 1 in original study DFA102, Week 52 was in extension study DFA102E. If Day 1 value was missing or after the first dose of drug, the last available value on or prior to Day 1 was used. Week 52, treatment stable evaluable population: those participants who enrolled and received at least 1 injection of any treatment (ITT); treatment regimens same in both DFA102/DFA102E (stable); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock).
Time Frame: Baseline (Day 1) to Week 52
Population: n=number of participants with non-missing data in each treatment group by test. glucose n=20,20,27,19; total cholesterol n=21,20,27,19; triglycerides n=21,20,27,19; LDL/HDL n=21,20,27,19. ITT population with treatment regimens same in DFA102/DFA102E (stable); completed Week 52; no major protocol deviations in DFA102 or DFA102E.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable
Number analyzed (Participants) | 21 | 20 | 27 | 19
mg/dL
  glucose | -1.88 [-5.62 to 1.85] | -0.60 [-4.36 to 3.17] | 0.03 [-3.38 to 3.43] | -6.29 [-10.07 to -2.50]
  total cholesterol | 4.19 [-8.25 to 16.63] | -2.21 [-15.10 to 10.68] | -3.24 [-14.84 to 8.35] | -3.84 [-17.12 to 9.43]
  triglycerides | -10.05 [-26.77 to 6.67] | -5.41 [-22.58 to 11.76] | -5.86 [-21.16 to 9.43] | -12.74 [-30.12 to 4.64]
  low density lipoprotein (LDL) | 13.43 [1.96 to 24.90] | 4.43 [-7.49 to 16.35] | 6.03 [-4.64 to 16.70] | 4.43 [-7.97 to 16.82]
  high density lipoprotein (HDL) | 2.92 [-0.36 to 6.21] | 7.96 [4.57 to 11.36] | 5.04 [2.01 to 8.08] | 7.61 [4.10 to 11.12]

7. Secondary Outcome: LS Mean Absolute Change From Baseline in Original Study DFA102 to Week 52 in Extension Study DFA102E in Total Insulin - Week 52 Evaluable Treatment Stable Population
Description: Total insulin was measured in micro international units per milliliter (µIU/mL). Baseline is Day 1 in original study DFA102. If Day 1 value was missing or after the first dose of drug, the last available value on or prior to Day 1 was used. Week 52, treatment stable evaluable population: those participants who enrolled and received at least 1 injection of any treatment (ITT); treatment regimens same in both DFA102/DFA102E (stable); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock).
Time Frame: Baseline to Week 52
Population: n=number of participants with non-missing data in each treatment group. ITT population (received at least 1 injection) with treatment regimens same in DFA102/DFA102E (stable treatment); completed Week 52; no major protocol deviations in DFA102/102E.
Measure: Least Squares Mean (95% Confidence Interval); unit: µIU/mL
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable
Number analyzed (Participants) | 21 | 19 | 25 | 18
µIU/mL | -0.54 [-2.97 to 1.89] | -2.16 [-4.71 to 0.39] | -0.62 [-2.94 to 1.70] | -1.61 [-4.20 to 0.97]

8. Secondary Outcome: Number of Participants Achieving at Least 5%, 10%, and 15% of Body Weight Loss From Original Study DFA102 Baseline to Week 52 in Extension Study DFA102E - Week 52 Evaluable Population
Description: Baseline is Day 1 in original study DFA102. If Day 1 value was missing or after the first dose of drug, the last available value on or prior to Day 1 was used. Percent change in body weight from baseline was categorized: Change greater than (>) 0% (Body weight gain); Change less than, equal to (<=) 0 to > -5% (No body weight change or body weight loss <5%); Change <= -5% (Body weight loss greater than, equal to (>=)5%); Change <= -5% to > -10% (Body weight loss >=5% and <10%); Change <= -10% (Body weight loss ≥10%); Change <= -10% to > -15% (Body weight loss >=10% and <15%); Change <= -15% (Body weight loss >=15%).
Time Frame: Baseline (Day 1) to Week 52
Population: Number analyzed with non-missing data at Week 52. Week 52 Evaluable Population: All ITT participants (received at least 1 injection);remained in the study through Week 52; complied with the protocol (per sponsor prior to database lock);no major deviations; some may have been excluded based on a clinical review of the data prior to database lock.
Measure: Number; unit: participants
Groups:
- 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 1.25 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 2.5 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 5.0 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono: Participants who received 5.0 mg metreleptin plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 5.0 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102. A blinded pramlintide dose escalation/titration in the first week of treatment was performed, to minimize nausea and/or vomiting.
Arm/Group | Placebo | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 27 | 19 | 12 | 7 | 6 | 20 | 29 | 30
participants
  Weight Loss >=5% and <10% | 3 | 4 | 10 | 6 | 6 | 1 | 1 | 6 | 7 | 7
  Weight Loss >=10% and <15% | 3 | 2 | 5 | 4 | 0 | 1 | 1 | 4 | 6 | 5
  Weight Loss >=5% | 8 | 12 | 21 | 12 | 7 | 3 | 4 | 15 | 18 | 18
  Weight Loss >=10% | 5 | 8 | 11 | 6 | 1 | 2 | 3 | 9 | 11 | 11
  Weight Loss >=15% | 2 | 6 | 6 | 2 | 1 | 1 | 2 | 5 | 5 | 6

9. Secondary Outcome: Number of Participants Achieving at Least 5%, 10% and 15% Body Weight Loss From Extension Study DFA102E Baseline (Week 28) to Week 52 - Week 52 Evaluable Population
Description: Baseline in extension study was Week 28; if value was missing or after the first dose in DFA102E, the last available value on or prior to Week 28 was used. Percent change in body weight from baseline was categorized: Change greater than (>) 0% (Body weight gain); Change less than, equal to (<=) 0 to > -5% (No body weight change or body weight loss <5%); Change <= -5% (Body weight loss greater than, equal to (>=)5%); Change <= -5% to > -10% (Body weight loss >=5% and <10%); Change <= -10% (Body weight loss ≥10%); Change <= -10% to > -15% (Body weight loss >=10% and <15%); Change <= -15% (Body weight loss >=15%).
Time Frame: Baseline (Week 28) to Week 52
Population: Participants analyzed had non-missing data at Week 52. Week 52 Evaluable Population: ITT participants (received at least 1 injection); remained in the study through Week 52; complied with the protocol (per sponsor prior to database lock); no major deviations; some may have been excluded based on a clinical review of the data prior to database lock.
Measure: Number; unit: participants
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 27 | 19 | 12 | 7 | 6 | 20 | 29 | 30
participants
  Weight Loss >=5% and <10% | 2 | 1 | 4 | 1 | 0 | 0 | 0 | 7 | 3 | 3
  Weight Loss >=10% and <15% | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
  Weight Loss >=5% | 2 | 3 | 4 | 1 | 0 | 0 | 2 | 8 | 3 | 5
  Weight Loss >=10% | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
  Weight Loss >=15% | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Mean Absolute Change From Original Study DFA102 Screening at Week 52 in Extension Study DFA102E in Susceptibility to Eating Questionnaire (SEQ) Item Scores - Week 52 Evaluable Population
Description: The eating questionnaire is an exploratory measure of appetite, satiety, and perceived control over portion size using 10 items, with each response measured on a 100 mm visual analogue scale (VAS). Ranges vary from: Never to Very Often; Not at All Difficult to Extremely Difficult; Not at all Strong to Very Strong). Lower scores show improvement. The Eating Questionnaire instructed participants to rate their responses to these items over the past 7 days. Values were obtained for this questionnaire on Visit 3 in the screening period in DFA102 and at Weeks 28, 40, and 52 in DFA102E.
Time Frame: Screening to Week 52
Population: Enrolled and received at least 1 injection of any treatment (ITT); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock); no major deviations during original study/extension. Additional exclusions based on clinical review of the data prior database lock.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono: Participants who received 5.0 mg metreleptin plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 5.0 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102.A blinded pramlintide dose escalation/titration in the first week of treatment was performed for participants who had not received 360 mcg pramlintide in DFA102, to minimize nausea and/or vomiting.
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 27 | 19 | 12 | 7 | 6 | 20 | 29 | 30
units on a scale
  Frequency of Food Cravings | -14.1 (16.91) | -14.4 (18.61) | -15.0 (23.59) | -21.4 (33.81) | -3.1 (19.21) | -22.6 (33.53) | -13.7 (41.94) | -18.9 (21.06) | -12.8 (21.82) | -21.4 (25.56)
  Strength of Food Cravings | -14.3 (15.48) | -13.3 (22.96) | -14.2 (22.26) | -17.9 (28.54) | 5.3 (19.35) | -30.3 (30.57) | -9.5 (32.57) | -13.0 (28.56) | -8.8 (25.08) | -14.6 (22.39)
  Difficult to Control Eating | -18.3 (25.17) | -19.7 (20.36) | -23.3 (27.38) | -17.6 (28.98) | -8.8 (19.64) | -31.6 (29.38) | -17.7 (27.47) | -22.1 (22.64) | -16.6 (24.54) | -28.7 (23.15)
  Difficult to Resist Food Cravings | -17.6 (25.36) | -20.0 (23.08) | -24.2 (25.77) | -16.9 (30.90) | -3.0 (20.43) | -30.9 (31.20) | -15.7 (36.47) | -25.6 (22.32) | -18.5 (23.65) | -25.8 (26.29)
  Eating in Response to Food Cravings | -18.4 (31.97) | -18.7 (26.60) | -20.4 (22.96) | -21.3 (30.83) | -1.8 (20.91) | -26.6 (32.46) | -7.3 (30.61) | -27.4 (17.41) | -13.4 (22.50) | -29.2 (26.61)
  Difficult to Control Portion Sizes | -24.6 (25.85) | -19.9 (21.13) | -25.0 (25.80) | -31.7 (30.85) | -6.6 (25.50) | -24.4 (26.68) | -11.5 (23.42) | -33.1 (20.46) | -24.4 (21.62) | -27.4 (24.34)
  How Hungry | -1.2 (20.40) | -12.8 (19.31) | -20.3 (23.23) | -12.9 (29.00) | 0.1 (25.54) | -17.9 (12.13) | -5.0 (20.61) | -20.8 (26.63) | -8.2 (25.80) | -16.2 (28.58)
  How Full After Meals | -6.5 (33.57) | -10.1 (22.03) | -1.9 (24.74) | 3.5 (29.96) | 0.8 (24.77) | -4.3 (44.84) | 11.8 (21.18) | -6.2 (23.42) | -1.3 (20.86) | -10.2 (27.99)
  Thoughts of Food | -8.5 (17.01) | -12.3 (16.06) | -17.9 (22.54) | -17.4 (32.05) | -1.5 (29.05) | -26.3 (22.97) | -14.5 (44.56) | -16.3 (22.70) | -6.0 (22.34) | -18.4 (24.90)
  How Pleasant Meals | -1.0 (17.16) | -2.8 (22.85) | 8.4 (24.09) | 15.5 (30.30) | 8.8 (21.84) | 8.4 (16.00) | 7.7 (13.09) | 7.1 (17.29) | 1.3 (20.91) | -5.2 (24.10)

11. Secondary Outcome: Mean Absolute Change From Original Study DFA102 Screening to Week 52 in Extension Study DFA102E in Binge Eating Scale (BES) Total Score - Week 52 Evaluable Population
Description: The Binge Eating Scale (BES) is a 16-item questionnaire that assesses the behavioral and cognitive correlates of binge eating, including participants' perceived self-control over eating behavior using a range of 1 to 4 with 1=positive perceptions and 4= negative perceptions. Lower scores show improvement. The minimum and maximum score for the BES instrument is 0 and 55, respectively; the higher the score the worse the outcome. Values were obtained for this questionnaire on Visit 3 in the screening period in DFA102 and at Weeks 28, 40, and 52 in DFA102E.
Time Frame: Screening to Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 27 | 19 | 12 | 7 | 6 | 20 | 29 | 30
units on a scale | -5.8 (7.09) | -5.7 (4.60) | -7.1 (7.31) | -7.4 (7.90) | -0.3 (7.98) | -10.4 (7.98) | -8.6 (2.41) | -8.1 (4.92) | -5.3 (7.97) | -8.1 (8.22)

12. Secondary Outcome: Mean Absolute Change From Original Study DFA102 Screening to Week 52 in Extension Study DFA102E in Hospital Anxiety and Depression Scale (HADS) Total Scores - Week 52 Evaluable Population
Description: The HADS is a questionnaire that uses 14 items to assess both anxiety and depression over the past week. The odd numbered items constitute the anxiety subscale, and the even numbered items constitute the depression subscale. The individual response scores for each subscale component are added together to obtain the individual subscale scores. The minimum and maximum score for each subscale is 0 and 21, respectively. Lower scores show improvement. Values were obtained for this questionnaire on Visit 3 in the screening period in DFA102 and at Weeks 28, 40, and 52 in DFA102E.
Time Frame: Screening to Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 31 | 35 | 36 | 28 | 13 | 14 | 13 | 29 | 37 | 37
units on a scale
  Change in Total Scores for Anxiety | -0.4 (2.94) | -1.2 (2.33) | -0.5 (2.84) | -0.2 (3.42) | -0.8 (3.31) | 0.1 (2.11) | 0.4 (1.43) | -0.7 (2.69) | -1.2 (3.45) | -0.8 (3.00)
  Change in Total Scores for Depression | -1.0 (3.46) | -2.1 (2.60) | -0.9 (1.70) | -0.3 (2.85) | 0.3 (2.66) | -1.0 (2.80) | -0.8 (2.44) | -1.3 (2.59) | -0.9 (2.26) | -1.7 (2.57)

13. Secondary Outcome: Mean Absolute Change From Original Study DFA102 Screening to Week 52 in Extension Study DFA102E in the Epworth Sleepiness Scale (ESS) Total Score - Week 52 Evaluable Population
Description: The Epworth Sleepiness Scale (ESS) is an eight-item questionnaire that assesses sleep propensity in daily situations of increasing sleepiness on a four-point scale with 0=would never doze and 3=high chance of dozing. Lower scores show improvement. Values were obtained for this questionnaire on Visit 3 in the screening period in DFA102 and at Weeks 28, 40, and 52 in DFA102E.
Time Frame: Screening to Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 27 | 19 | 12 | 7 | 6 | 20 | 29 | 30
units on a scale | -2.0 (4.52) | -2.5 (3.17) | -2.5 (3.13) | -1.3 (3.28) | 0.2 (4.41) | -3.9 (3.18) | 0.0 (1.67) | -1.3 (3.34) | -1.2 (2.42) | -1.1 (4.15)

14. Secondary Outcome: Total Trough Concentration of Plasma Leptin at Baseline and at Weeks 40, 52, and End of Treatment Follow up - Week 52 Stable Evaluable Population
Description: Mean fasting plasma total leptin concentration (nanograms per milliliter; ng/mL) change from baseline over time by pooled metreleptin dose (sex, baseline BMI category, and baseline value). Baseline defined as Day 1 in DFA102 study and Week 28 in study DFA102E. If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Follow up occurred 3-28 days after end of treatment. Leptin concentrations were measured using a validated immunoenzymetric assay utilizing polyclonal capture antibody, monoclonal detection antibody, and colorimetric readout by Amylin Pharmaceuticals, Inc. Week 52 Stable Evaluable: Enrolled and received at least 1 injection of any treatment (ITT); treatment regimens same in both DFA102/DFA102E (stable); evaluable: completed Week 52; complied with protocol, (per Sponsor prior to database lock); no major deviations during original study/extension.
Time Frame: Baseline to end of treatment follow up
Population: number (n) of participants who are Week 52 evaluable in a stable treatment sequence (received the same treatment in both DFA102 and DFA102E) and who had follow up data. Week 52 in Metreleptin 2.5 mg arm n=55 (all others n=56); Week 40 in Metreleptin 5 mg arm n=66 (all others n=68)
Measure: Geometric Mean (Standard Error); unit: ng/mL
Groups:
- Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 1.25 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E.
- Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 2.5 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E.
- Pramlintide 360 Mcg + Metreleptin 5 mg - Stable: Pramlintide 360 mcg BID plus Metreleptin 5 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E.
Arm/Group | Pramlintide 360 Mcg + Metreleptin 1.25 mg - Stable | Pramlintide 360 Mcg + Metreleptin 2.5 mg - Stable | Pramlintide 360 Mcg + Metreleptin 5 mg - Stable
Number analyzed (Participants) | 20 | 56 | 68
ng/mL
  Baseline in DFA102 (Day 1) | 32.50 (4.990) | 34.48 (3.089) | 29.50 (2.251)
  Baseline in DFA102E (Week 28) | 102.02 (17.466) | 232.48 (29.371) | 420.24 (48.012)
  Week 40 | 96.23 (19.418) | 236.02 (29.856) | 416.52 (58.352)
  Week 52 | 88.47 (17.576) | 177.32 (25.765) | 259.85 (40.650)
  Follow up after end of treatment | 52.90 (9.584) | 89.21 (11.180) | 89.49 (11.712)

15. Secondary Outcome: Mean Change in Systolic and Diastolic Blood Pressure From Baseline of DFA102 at Week 52 of DFA102E - Intent to Treat Population
Description: Baseline refers to Day 1 of original study DFA102. If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Blood pressure was taken while the participant was sitting and was measured in millimeters of mercury (mm Hg).
Time Frame: Baseline (Day 1) to Week 52
Population: Enrolled and received at least 1 injection of any treatment; had data available.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- 360 mcg Pramlintide + 1.25mg Metreleptin - Stable: Pramlintide 360 mcg BID plus Metreleptin 1.25 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
- 360 mcg Pramlintide + 2.5 Metreleptin - Stable: Pramlintide 360 mcg BID plus Metreleptin 2.5 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
- 360 mcg Pramlintide + 5.0 Metreleptin - Stable: Pramlintide 360 mcg BID plus Metreleptin 5.0 mg BID self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 28 | 22 | 12 | 7 | 8 | 20 | 31 | 30
mm Hg
  Systolic Blood Pressure | -1.0 (9.91) | 1.8 (12.74) | -4.6 (14.54) | -4.9 (10.88) | 0.7 (14.57) | 3.7 (14.35) | -6.4 (6.21) | -2.9 (9.75) | -7.0 (9.63) | -4.8 (10.94)
  Diastolic Blood Pressure | -0.6 (5.40) | -0.6 (9.17) | -2.7 (7.29) | -1.5 (9.98) | -1.7 (8.56) | -0.3 (7.74) | -5.3 (8.94) | -5.8 (8.17) | -2.5 (9.77) | -4.0 (5.99)

16. Secondary Outcome: Mean Change in Heart Rate From Baseline of DFA102 at Week 52 of DFA102E - Intent to Treat Population
Description: Baseline refers to Day 1 of original study DFA102. If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Heart rate was measured while the participant was sitting and was measured in beats per minute (bpm).
Time Frame: Baseline to Week 52
Population: Enrolled and received at least 1 injection of any treatment; had data available.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 28 | 22 | 12 | 7 | 8 | 20 | 31 | 30
bpm | -3.1 (9.22) | -1.8 (9.39) | -3.1 (6.49) | -1.4 (7.73) | -1.6 (5.81) | 0.9 (9.25) | -0.9 (11.75) | -2.6 (8.39) | -4.0 (7.12) | -2.8 (6.58)

17. Secondary Outcome: Mean Change From DFA102 Screening at Week 52 in Study DFA102E for Electrocardiogram Parameters - Intent to Treat Population
Description: A 12-Lead electrocardiogram (ECG) was obtained. The PR interval, which is the time from beginning of the P wave to the beginning of the QRS complex (Note: QRS complex is a name for the combination of 3 of the graphical deflections seen in an ECG); QRS interval, which is time from the beginning to the end of the QRS complex; QT interval (measure between Q wave and T wave in the heart's electrical cycle); and QT interval corrected for heart rate using Fridericia's formula (QTcF) were measured in milliseconds (msec).
Time Frame: Screening to Week 52
Population: Enrolled and received at least 1 injection of any treatment; had ECG data available at Week 52.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 28 | 21 | 12 | 7 | 8 | 19 | 31 | 30
msec
  PR Interval | 1.2 (10.29) | 1.2 (22.15) | 3.6 (14.11) | 0.6 (13.14) | 15.8 (52.77) | 6.0 (8.49) | 2.5 (9.50) | -2.3 (10.83) | 1.8 (13.80) | 0.9 (10.82)
  QRS | -0.2 (5.19) | 3.4 (11.05) | 1.8 (6.81) | 1.0 (5.76) | -2.4 (14.09) | 1.6 (4.24) | 0.0 (9.56) | 1.7 (5.50) | 0.5 (6.15) | -0.9 (4.35)
  QT Interval | 15.3 (28.67) | 8.1 (32.50) | 15.6 (22.54) | 8.2 (26.37) | 19.4 (18.57) | 13.3 (25.00) | 2.5 (23.10) | 14.4 (31.39) | 5.5 (20.21) | 16.7 (16.94)
  QTcF | 1.3 (22.08) | 0.3 (16.64) | 1.4 (16.69) | -2.2 (18.96) | 7.1 (11.66) | 5.1 (24.22) | 6.5 (15.19) | 3.2 (24.49) | -1.7 (16.34) | 0.8 (16.23)

18. Secondary Outcome: Number of Hematology or Urinalysis Laboratory Values of Potential Clinical Importance Observed From Baseline of DFA102E to Week 52 - Intent to Treat Population
Description: Baseline defined as Week 28 (first week of study DFA102E). Hematology: Hematocrit males <36%, females <30%. Hemoglobin males <12 g/dL, females <10 g/dL. White blood cell count (WBC) H >18,000/µL; L <1,500/µL. Urinalysis: Urine protein H >= 3+ or >= 500 mg/dL. Urine glucose H >= 3+ or >= 500 mg/dL. Urine ketones >= 3+ or Large. Laboratory values were obtained at Weeks 28, 36, 44, and 52. Numbers of values are cumulative across the extension
Time Frame: Baseline to Week 52
Population: Enrolled and received at least 1 injection of any treatment; participants had laboratory data available; platelet counts: n=19 in second arm (not 20); n=20 in fourth arm (not 22); n=11 in fifth arm (not 12);
Measure: Number; unit: number of laboratory values
Groups:
- 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram: Participants who received 180 mcg pramlintide plus 5.0 mg metreleptin self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg pramlintide plus 5.0 mg metreleptin in the extension study for up to 52 Weeks, inclusive of DFA102.A blinded pramlintide dose escalation/titration in the first week of treatment was performed for participants who received 180 mcg pramlintide in DFA102, to minimize nausea and/or vomiting.
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 20 | 20 | 27 | 22 | 12 | 7 | 8 | 20 | 31 | 30
number of laboratory values
  Hematocrit | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Chemistry Laboratory Values of Potential Clinical Importance Observed From DFA102E Baseline to Week 52 - Intent to Treat Population
Description: Baseline defined in study DFA102E as Week 28. Criteria for laboratory values of potential clinical importance for obese and overweight (BMI>=25 kg/m^2) participants: Total bilirubin High (H) > 2 mg/dL; Plasma or serum glucose fasting or non-fasting H > 200 mg/dL, low (L) < 60 mg/dL; Albumin L <2.5 g/dL; Creatine kinase H > 3*Upper limit of Normal (ULN); Sodium L <130 milliequivalents per liter (mEq/L), H > 150 mEq/L; potassium L<3.0 mEq/L, H> 5.5 mEq/L;bicarbonate L<18 mEq/L, H>35 mEq/L;calcium L <8mg/dL, H> 11 mg/dL; triglycerides H> 500 mg/dL; Cholesterol L < 100 mg/dL, H > 350 mg/dL; Alkaline phosphatase H > 3*ULN; Gamma-glutamyltransferase H>3*ULN; creatinine males > 1.6 mg/dL, females > 1.4 mg/dL; alanine aminotransferase H > 3*ULN; aspartate aminotransferase H > 3*ULN; urea nitrogen H > 45 mg/dL; uric acid males > 10.0 mg/dL, females > 8.0 mg/dL; Phosphorus L < 1.0 mg/dL H > 6.0 mg/dL. Laboratory values obtained at Weeks 28, 36, 44, and 52; number of values a
Time Frame: Baseline to Week 52
Population: All Enrolled participants who received at least one injection of any study medication in Study DFA102E; had laboratory data available. Number analyzed presented above is at Week 52; Number analyzed at Week 28: N= 31, 35, 36, 28, 13, 14, 13, 29, 37, 37.
Measure: Number; unit: Number of Laboratory values
Groups:
- 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram: Participants who received 180 mcg pramlintide plus 2.5 mg metreleptin self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg pramlintide plus 2.5 mg metreleptin in the extension study for up to 52 Weeks, inclusive of DFA102.A blinded pramlintide dose escalation/titration in the first week of treatment was performed for participants who received 180 mcg pramlintide in DFA102, to minimize nausea and/or vomiting.
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Number analyzed (Participants) | 21 | 20 | 28 | 22 | 12 | 7 | 8 | 20 | 31 | 30
Number of Laboratory values
  alanine aminotransferase (ALT) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Bicarbonate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Creatine kinase | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Calcium | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
  Creatinine | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma-glutamyltransferase | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
  Potassium | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Uric Acid | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 3 | 2

20. Secondary Outcome: Number of Participants With Treatment Emergent Positive Anti-leptin Antibody Titers at Week 52 and at Follow up by Metreleptin Dose - Intent to Treat Population
Description: Baseline refers to Day 1. If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Follow up occurred on Days 3 - 28 after treatment ended. Serum titer determinations for antibodies to metreleptin were made using a validated electrochemical luminescence (ECLA) bridging assay. Antibody titers were assessed according to the following dilutions: 0, 5, 25, 125, 625, 3125, 15625, and 78125. Participants were considered to have a positive titer to treatment-emergent antibodies to metreleptin at a given visit if they had a titer >=5 following a negative or missing titer at baseline or if they had a titer that had increased by at least 2 dilutions from a detectable level at baseline.
Time Frame: Baseline to end of treatment follow up
Population: N for Week 52 presented above. For Follow up: N=18,58,68,11,7,8.
Measure: Number; unit: participants
Groups:
- 360 mcg Pramlintide + Metreleptin 1.25 mg - Stable: Participants who received 360 mcg pramlintide plus 1.25 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
- 360 mcg Pramlintide + Metreleptin 2.5 mg - Stable: Participants who received 360 mcg pramlintide plus 2.5 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
- 360 mcg Pramlintide + Metreleptin 5 mg - Stable: Participants who received 360 mcg pramlintide plus 5.0 mg metreleptin self administered SC for up to 52 Weeks, inclusive of DFA102.
  Stable: same treatment regimen in both DFA102 and DFA102E
- 360 mcg Pramlintide + Metreleptin 1.25 mg - Prior Monotherapy: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 1.25 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + Metreleptin 2.5 mg - Prior Monotherapy: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 2.5 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102.
- 360 mcg Pramlintide + Metreleptin 5 mg - Prior Monotherapy: Participants who received 360 mcg pramlintide plus placebo (monotherapy) self administered SC in the original study DFA102, and who consented to enter the extension study DFA102E, were treated with 360 mcg Pramlintide plus 5.0 metreleptin in this group of the extension study, for up to 52 Weeks, inclusive of DFA102.
Arm/Group | 360 mcg Pramlintide + Metreleptin 1.25 mg - Stable | 360 mcg Pramlintide + Metreleptin 2.5 mg - Stable | 360 mcg Pramlintide + Metreleptin 5 mg - Stable | 360 mcg Pramlintide + Metreleptin 1.25 mg - Prior Monotherapy | 360 mcg Pramlintide + Metreleptin 2.5 mg - Prior Monotherapy | 360 mcg Pramlintide + Metreleptin 5 mg - Prior Monotherapy
Number analyzed (Participants) | 20 | 58 | 71 | 12 | 7 | 8
participants
  Week 52 | 20 | 58 | 71 | 8 | 7 | 7
  Follow up after end of treatment | 17 | 57 | 68 | 8 | 7 | 7

ADVERSE EVENTS:
Time Frame: 52 Weeks, intent to treat population. Enrolled and treated with at least one injection during the extension study DFA102E.
Arm/Group | Placebo - Stable | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable | 360 mcg Pramlintide + 2.5 Metreleptin - Stable | 360 mcg Pramlintide + 5.0 Metreleptin - Stable | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35 | 0/36 | 0/28 | 0/13 | 0/14 | 0/13 | 2/29 | 1/37 | 1/37
Other Adverse Events (participants affected / at risk) | 20/31 | 25/35 | 29/36 | 19/28 | 10/13 | 11/14 | 12/13 | 26/29 | 28/37 | 28/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Stable (N=31) | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable (N=35) | 360 mcg Pramlintide + 2.5 Metreleptin - Stable (N=36) | 360 mcg Pramlintide + 5.0 Metreleptin - Stable (N=28) | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 (N=13) | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 (N=14) | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 (N=13) | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono (N=29) | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram (N=37) | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram (N=37)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Stable (N=31) | 360 mcg Pramlintide + 1.25mg Metreleptin - Stable (N=35) | 360 mcg Pramlintide + 2.5 Metreleptin - Stable (N=36) | 360 mcg Pramlintide + 5.0 Metreleptin - Stable (N=28) | 360 mcg Pramlintide + 1.25 mg Metreleptin - Prior Mono+1.25 (N=13) | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Mono+2.5 (N=14) | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Mono+5.0 (N=13) | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Metre Mono (N=29) | 360 mcg Pramlintide + 2.5 mg Metreleptin - Prior Lower Pram (N=37) | 360 mcg Pramlintide + 5.0 mg Metreleptin - Prior Lower Pram (N=37)
nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 11 (13) | 7 (9) | 8 (12)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 5 (8) | 7 (7) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 7/12 (8)
sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 6 (6) | 4 (5)
nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 5 (6) | 3 (3) | 0 (0)
injection site hemorrhage (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 4 (4)
injection site bruising (General disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (3) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
headache (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (4)
injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
injection site nodule (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
gastroenteritis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
injection site erythema (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (2)
anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3)
ear infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
back injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
injection site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
edema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
aphthous stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
enteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
tooth abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
conjunctival edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypoesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.